CLINICAL TRIAL: NCT03389581
Title: The Effect of Awareness on Preoperative Anxiety Before Anesthesia
Brief Title: The Effect of Awareness on Preoperative Anxiety
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: awareness
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Anxiety; Anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: awareness and anxiety — before operation awareness and anxiety will recorded with STAIX-I score

SUMMARY:
In the majority of patients, anxiety and fear are observed at different levels before surgery. Preoperative anxiety was reported in 60-80% of the patients who underwent surgery. This anxiety and fear can be attributed to many factors. Some of these are mainly anesthesia, previous experience of the patient, personality traits, concerns about surgical intervention, and postoperative pain. Patients' anxiety levels can be influenced by a variety of factors, including previous experience, type of hospital arrival, sex, age, and type of surgery.Anesthesia-related awareness among the experiences of anesthesia is described in the literature. In a study of 20,402 patients in the United States, the awareness rate was 0.13%. Being aware is that the patient is awake during the surgery and recalls seeing bad dreams. At that time the patient could not specify this because he was immobile. Being awake is that the patient is awake and showing it through his movements. The patient may not remember this situation later. It is a condition that can always be overlooked in previous experience, which is an important parameter of anxiety in the preoperative period. The patients included in the study were planned to use the modified Brice awareness score, first mentioned in 1970 as the name of the person who used the anesthesia and anesthesia for awareness. In this study, investigators aim to reveal the effect of anesthesia awareness on preoperative anxiety in patients with previous anesthesia story.

DETAILED DESCRIPTION:
in this study will include 300 patients. 300 patients will be enrolled in the anesthesia outpatient clinic scheduled for elective surgery for any reason at the age of 18-65 years. Patients with dementia and psychiatric disorders, anxiolytic and psychiatric drug users and patients who can not receive written approval will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* all patients between 18-70 yr

Exclusion Criteria:

* dementia
* psychiatric disorders
* using antipsychotic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-70
Study Population: elective surgery for any reason
Sampling Method: Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
awareness | preoperative visit before surgery
  modify Brice Score

SECONDARY OUTCOMES:
anxiety | preoperative visit before general anesthesia
  The State and Trait Anxiety Inventory (STAI-S) score will used

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Siences Diskapi Yildirim Beyazit T&R hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided